CLINICAL TRIAL: NCT03618186
Title: Neuroimaging Study
Status: Enrolling by invitation | Phase: Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Neill R. Graff-Radford, M.D., Principal Investigator, Mayo Clinic
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-008710; 5P50AG016574-20 (NIH)
Record Dates: First submitted 2018-08-02; First posted 2018-08-07 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Cognitive Impairment
Keywords: African Americans; neurological exam; Dementia; Alzheimer's Disease
MeSH Terms: conditions — Cognitive Dysfunction; Dementia; Alzheimer Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Normal control (Experimental): Cognitively normal volunteers
  Interventions: Combination Product: Tau PET scan
- Mild Cogntive impairment (Experimental): Person with cognitive impairment that meet Peterson Criteria
  Interventions: Combination Product: Tau PET scan
- Demented (Experimental): Patient's that meet dementia criteria
  Interventions: Combination Product: Tau PET scan

INTERVENTIONS:
Combination Product: Tau PET scan — Patient will receive a dose of flutaucipir and be scanned appropriately

SUMMARY:
The researchers are trying to gather information and learn more about imaging tests in racially different people who are cognitively normal or have dementia.

ELIGIBILITY:
Inclusion Criteria:

* Male or female African Americans 30 years of age or older
* Subjects who have completed or are scheduled to undergo the neurological evaluation procedures described below.

Exclusion Criteria:

* Subjects unable to lie down without moving for 20 minutes.
* Women who are pregnant or cannot stop breast feeding for 24 hours.
* Claustrophobic patients unable to tolerate the scans.
* Subjects with a prolonged QT interval (as demonstrated by ECG test) cannot participate in the Tau-PET scans.
* Standard safety exclusionary criteria for MRI such as metallic foreign bodies, pacemaker, etc, since the quantitative PET data analysis is based on anatomic criteria that are established uniquely for each subject by registration to his/her MRI.

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2018-11-26 (Actual); Primary Completion 2030-05 (Estimated); Study Completion 2030-05 (Estimated)

PRIMARY OUTCOMES:
Tau positive scans | 5 years
  Percentage of each of the three groups with tau positive scans

CONTACTS AND LOCATIONS:
Overall Officials: Neill R Graff-Radford, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic Minnesota, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: No